CLINICAL TRIAL: NCT06080139
Title: A Community-based Participatory Study to Support Parenting and Improve Family Mental Health in Refugee Shelters in Tijuana, Mexico
Brief Title: Supporting Refugee Parenting Community and Family Mental Health in Tijuana
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Universidad Iberoamericana (Other); PILA Global (Unknown); Fulbright (Other)
Responsible Party: Principal Investigator, Xinshu She, MD, MPH, Clinical Associate Professor of Pediatrics, Stanford University
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: 69854
Record Dates: First submitted 2023-08-22; First posted 2023-10-12 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Refugee Health
Keywords: parenting; parental mental health; child behavior; prevention
MeSH Terms: conditions — Child Behavior

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- parenting sessions group (Experimental): This arm will receive a culturally adapted parenting curriculum twice a week for 4 weeks during month 3 of the study
  Interventions: Behavioral: Refugee parenting education in a participatory community
- waitlist control group (Active Comparator): This arm will receive a handout about parenting techniques in Spanish during month 3. They then receive the same parenting curriculum during month 4.
  Interventions: Behavioral: Refugee parenting education in a participatory community

INTERVENTIONS:
Behavioral: Refugee parenting education in a participatory community — Parents will vote for one of the 5 previously studied refugee parenting curriculums: 1) Creating Opportunities Through Mentoring Parenting Involvement and Safe Space (COMPASS); 2) GenerationPMTO; 3) Happy Families; 4) Family Strengthening Intervention for Refugees (FSI-R).
  Researchers will use a model of Learning by Observing and Pitching In (LOPI), to empower community members in the learning process. LOPI is a multicomponent way of organizing group learning that improves collaboration, alertness, and executive functions such as perspective-taking and self-regulation in addition to specific skills learning and has been used in many indigenous and indigenous-heritage communities of the Americas.

SUMMARY:
The goal of this study is to better understand and support parenting practices and family mental health among migrant parents in Tijuana, Mexico. the main questions it aims to answer are:

1. What parenting skills are most needed for learning?
2. How can we teach them in a participatory way respecting cultural values and norms?
3. How does this parenting program affect parental and child interactions and mental health?

Participants will

1. have the opportunity to give their opinions on the priority parenting skills needed and on which curriculum to use for learning these skills;
2. participate in small group learning sessions twice a week for 4 weeks;
3. be asked to complete a few surveys before and after the learning sessions, and 2 months after they complete the learning sessions.

Researchers will compare parents randomly assigned to parenting sessions group with waitlist control group (starting learning sessions 1 month later) to see if the group learning benefits parent-child interactions, parental stress, and parental confidence in parenting.

DETAILED DESCRIPTION:
Month 1:

The researchers will use a participatory research model to convene focus groups engaging community stakeholders in two large shelters in Tijuana to prioritize 3-5 parenting skills.

Month 2:

The researchers will recruit participating parents until reaching a sample size of 120, divided into 8 groups of 15. All participants will vote for 1-2 interventions from a list of 5 to revise and adapt to the local context through small group discussions and consensus building.

Month 3:

Participants will complete baseline questionnaires anonymously. Half of the participants (Group 1, N=60) will be randomized to receive the adapted learning curriculum in groups of 15, twice a week for 4 weeks. At the conclusion of month 3, all participants will complete the same questionnaires as pre-intervention. These data will serve as post-intervention data for Group 1 and a second baseline for the remaining participants (Group 2). During month 3, Group 2 will receive a two-page handout on childhood nutrition in Spanish. They will serve as the "control group" for the first wave of intervention.

Month 4:

Group 2 will receive the same intervention as group 1 in month 3. At the conclusion of month 4, participants will complete the same questionnaires as pre-intervention. They will also complete open-ended feedback interviews.

Month 5:

Researchers will analyze all anonymous data and share preliminary results with the community through peer leaders.

Month 6-7:

Researchers will conduct a phone follow-up for all available participants (2 months post intervention) and collect data anonymously.

Month 8:

Researchers will again analyze the aggregate data and share results with the community.

Month 9:

Researchers will draft a manuscript, share final results with the community and nonprofit/academic partners.

ELIGIBILITY:
Inclusion Criteria:

* all consenting parents staying at refugee shelters in Tijuana

Exclusion Criteria:

* known date of leaving Tijuana in less than 3 months

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2024-02-06 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-06-23 (Actual)

PRIMARY OUTCOMES:
parenting knowledge | immediately before intervention and after 4-week intervention period
  20 multiple choice questions (scores 0-20)
Child behavior and parental efficacy | immediately before intervention and after 4-week intervention period
  Child Adjustment and Parent Efficacy Scale (total scores 0-81, parental efficacy scores 19-190)

SECONDARY OUTCOMES:
Observed parent-child interactions | immediately before intervention, after 4-week intervention period, and 2-month post-intervenion follow-up
  Parenting Interactions with Children: Checklist of Observations Linked to Outcomes
parental stress | immediately before intervention, after 4-week intervention period, and 2-month post-intervenion follow-up
  Parent Stress Index-Short Form21
Qualitative feedback | after 4-week intervention period and at 2-month post-intervenion follow-up
  semi-structure interviews on program feedback and future suggestions
parenting knowledge | post intervention and at 2-month post-intervenion follow-up
  20 multiple choice questions (scores 0-20)
Child behavior and parental efficacy | post interventionand and at 2-month post-intervenion follow-up
  Child Adjustment and Parent Efficacy Scale (total scores 0-81, parental efficacy scores 19-190)

CONTACTS AND LOCATIONS:
Overall Officials: Xinshu She, MD, MPH, Principal Investigator — Stanford University
Locations (1):
- Canyon Nest, Tijuana, Estado de Baja California, Mexico

IPD SHARING:
Plan to Share IPD: No
There will be no individual data after completion of the data collection. All data will be anonymous and analyzed as collective data.

REFERENCES:
- See also: Stanford link to study description and contact — https://globalhealth.stanford.edu/programs/a-community-based-participatory-study-to-support-parenting-and-improve-family-mental-health-in-refugee-shelters-in-tijuana-mexico/